CLINICAL TRIAL: NCT05964309
Title: Effect of Preoxygenation in Sitting Position on The Oxygen Reserve Index (ORI) Alarm Time as Early Predictor of Impending Hypoxemia During Prolonged Apnea
Brief Title: Pre-oxygenation in Sitting Position and Oxygen Reserve Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Roshdi R Almetwalli, Professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-2022-01-446
Record Dates: First submitted 2023-06-11; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hypoxemia
Keywords: Oxygen reserve index; Preoxygenation; Hypoxemia; Sitting position
MeSH Terms: conditions — Hypoxia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine group(Control group) (Experimental): Supine group (flat head position- n=28) during pre-oxygenation patients will be in supine position
  Interventions: Other: supine group
- sitting group (Experimental): Sitting position (90 degree head up position- n=28) during pre-oxygenation patients will be in 90 degree head up position
  Interventions: Other: sitting group

INTERVENTIONS:
Other: supine group — after pre-oxygenation in supine position general anesthesia will be established then apnea alarm time will be recorded and compared with other group
  Other Names: control group
  Arms: Supine group(Control group)
Other: sitting group — after pre-oxygenation in sitting position general anesthesia will be established then apnea alarm time will be recorded and compared with other group
  Arms: sitting group

SUMMARY:
This prospective, controlled and randomized study aims at comparing the effect of position on the oxygen reserve index alarm time which is considered as predictor of hypoxemia in prolonged apnea which might be faced during general anesthesia (GA) in several situations such as the time from induction of anesthesia till endotracheal intubation.

participants will be divided into two groups; supine (n=38) and sitting group (n=38) both group will undergo elective procedures under GA and endotracheal intubation

DETAILED DESCRIPTION:
Introduction Pre oxygenation with high fraction of inspired oxygen is not only recommended before anesthesia induction and intubation but also to delay apnea induced hypoxemia in a variety of airway management and patients with limited oxygen reserve. As well as, to prolong the duration of apneic oxygenation in some airway interventions. Several methods have been used to improve the efficiency of pre oxygenation with controversial outcome. One of these methods is the performance of pre oxygenation in head up position.

During anesthetic management, pulse oximeter has been considered as valuable noninvasive tool for monitoring of patient oxygen saturation (SpO2%).

However, the relationship between the oxygen saturation (SpO2%) and the arterial partial pressure of oxygen (PaO2) restricts the pulse oximeter monitoring of patient oxygenation due to the sigmoidal pattern of this relation, as small changes only in SpO2% occur with increase in arterial oxygen tension above 80 mmHg., Therefore, when oxygen is provided, SpO2 remains 100% over a wide range of PaO2 (>80 mmHg) So It does not reflect the degree of hyperoxia during oxygen supplementation. On the other hand, when PaO2 is falling, the SpO2 may remain 100% until the PaO2 falls below approximately 80 mm Hg. Thus, it does not predict the onset of hypoxia in an apneic patient.

Oxygen reserve index (ORI) is a non-invasive real time non-unit scale between 0.00 and 1.00, which reflects the level of venous blood oxygen saturation (SvO2). When the patient is breathing room air ORI is 0.00, With oxygen supplementation, after SpO2 reaches its plateau of 100%, SvO2 continues rising as PaO2 increasing, and at PaO2 200mmHg usually ORI reaches a plateau. Hence ORI will serve to indicate PaO2 trends (rising or falling) in the range of 100-200 mmHg), so it will reflect the range of moderate hyperoxia (PaO2 ranging from 100 to 200 mmHg) during oxygen supply and, on the other hand, it will predict impending desaturation ahead of standard pulse oximetry during safe prolonged apnea technique in surgical patients at high risk.

Our study aims at assessment of the effect of pre oxygenation in sitting position on the ORI warning time for impending de-saturation during safe prolonged apnea techniques.

Methodology After approval of Institution Review Board and obtaining written informed consent from all participants, this prospective randomized controlled study will be conducted at King Fahd University hospital. Written, informed consent will be obtained from 56 illegible participants scheduled for elective surgery with planned general anesthesia with endotracheal intubation and invasive blood pressure monitoring (arterial line).

According to the head position during pre-oxygenation, participants will be randomly allocated via a computer-generated sequence into two groups; supine group (flat head position- n=28) and sitting group (90 degree head up position- n=28).

In the operation room standard monitoring will be applied. ORI sensor (Masimo RD lite) will be attached to the participant finger.

After recording the baseline vital signs, pre oxygenation in the three groups will be started by asking participants to spontaneously breath 100% oxygen via a well fitted face mask for 3 minutes, with rising of end-tidal fraction of oxygen (EtO2) to at least 0.9 and/or ORI to a plateau value. Rapid sequence induction and intubation using fentanyl, propofol, and succinylcholine will be performed with the aid of video assisted laryngoscope. The appropriate position of the endotracheal tube will be confirmed with direct vision and, will be disconnected from the breathing circuit (to prevent oxygenation while the patient is apneic) and exposed to the room air until SpO2 decreased to 94% then tube will be connected to the breathing circuit. Thereafter ventilator setting and anesthetic management will be according to the decision of the anesthesiologist assigned for patient care at this operative theater. ORI, SpO2 and PaO2 data were measured at four specific times (1) baseline (2) at the end of pre-oxygenation (3) at ORI alarm (4) when SpO2 reached 94%. The participant will be excluded from the study if he has failed pre oxygenation (EtO2 < 0.9 and/or ORI does not reach a plateau value after 3 min. pre oxygenation.

Statistical analysis If the difference between the mean ORI alarm time in the sitting group and the supine group is assumed to be 25 seconds, and a pooled standard deviation of 33 seconds., 28 participants in each group with a total of 56 participant would be an appropriate sample size to provide a significance of 5% and a power of 80%.

Data that will be normally distributed will be compared using t-test. Whereas Mann-Whitney test will be used to compare data with abnormal distribution. Fisher's exact test or Chi square test will be used to compare categorical data or gender ratio. Probability (p-value) less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Age 18-60 years
* General Anesthesia with endotracheal intubation

Exclusion Criteria:

* Significant cardiac or pulmonary disease.
* Anticipated difficult intubation.
* History of seizures.
* BMI 30kg/m2 or more.
* Smoking.
* Anemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Oxygen reserve index (ORI)alarming time | baseline, immediately after intubation, ORI warning alarm
  time from intubation till ORI alarm in minutes

SECONDARY OUTCOMES:
safe apnea time | baseline, immediately after intubation, when SpO2 % drop to 94% assessed in first 10 minutes after induction of general anesthesia
  time from intubation till Oxygen saturation (SpO2) drop to 94%.
Maximum Oxygen Reserve | Baseline, immediately after preoxygenation
  arterial oxygen tension (PaO2) after completion of pre-oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- King Fahd University Hospital, Khobar, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No